CLINICAL TRIAL: NCT01868477
Title: An Open-label, Phase II, Randomized, Pilot Study to Assess the Effect in Term of Erythroid Improvement of Deferasirox Combined With Erythropoietin Compared to Erythropoietin Alone in Patients With low-and Int-1-risk Myelodysplastic Syndrome.
Brief Title: Combination Study of Deferasirox and Erythropoietin in Patients With Low- and Int-1-risk Myelodysplastic Syndrome.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CICL670A2421
Record Dates: First submitted 2013-05-30; First posted 2013-06-04 (Estimated); Results first posted 2018-10-31 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Low and Int 1-risk Myelodysplastic Syndrome
Keywords: myelodysplastic syndrome; MDS; myelodysplasia; blood disorder; cytopenias; low blood counts; progressive bone marrow failure; adult; ICL570; deferasirox; erythropoietin; erythropoiesis; NF-kB pathway; hematopoiesis.
MeSH Terms: conditions — Myelodysplastic Syndromes; Anemia, Refractory, with Excess of Blasts; Hematologic Diseases; Cytopenia | interventions — Deferasirox; Epoetin Alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Erythropoietin alpha (Experimental): Patients will receive erythropoietin 40,000 units/week. If after 4 weeks erythroid improvement is inadequate, dose will be escalated to 60,000 units/week. If after 12 weeks of treatment, erythroid improvement in inadequate, patients will be switched to the combination arm. At any time when erythroid response is achieved, erythropoietin treatment will be stopped until end of study.
  Interventions: Drug: Erythropoietin alpha
- Deferasirox + Erythropoietin alpha (Experimental): Patients will receive deferasirox dispersible tablet (DT) 10 mg/kg/day or deferasirox film-coated tablet (FCT) 7 mg/kg/day in combination with erythropoietin 40,000 units/week. If after 4 weeks erythroid improvement is inadequate, erythropoietin dose will be escalated to 60,000 units/week. If after 12 weeks of treatment, erythroid improvement in inadequate, patients will be discontinued from the study. At any time when erythroid response is achieved, erythropoietin treatment will be stopped until end of study. Patients will continue deferasirox treatment.
  Interventions: Drug: Deferasirox DFX, DT; Drug: Deferasirox DFX, FCT

INTERVENTIONS:
Drug: Deferasirox DFX, DT — provided as dispersible tablets for oral use in 125 and 250, 500 mg
  Arms: Deferasirox + Erythropoietin alpha
Drug: Erythropoietin alpha
  Arms: Erythropoietin alpha
Drug: Deferasirox DFX, FCT — provided as film-coated tablet for oral use in 90, 180, 360 mg strengths
  Arms: Deferasirox + Erythropoietin alpha

SUMMARY:
The primary purpose of this trial was is to assess the effect of treatment with deferasirox combined with erythropoietin vs. erythropoietin alone on erythropoiesis in patients with low- and int-1-risk myelodysplastic syndrome. The addition of deferasirox to erythropoietin can lead to a potential synergism with the reduction of reactive oxygen species, through both the NF-kB pathway and the control of free toxic iron. This may create a better environment in the bone marrow for a better response with erythropoietin.

This study was designed to test in a prospective way the combination of deferasirox with erythropoietin in terms of their effect on hematopoiesis.

DETAILED DESCRIPTION:
This study did not meet the original enrollment objective of 60 patients and was terminated without extending enrollment past original planned LPFV of 31-Oct-2016.

ELIGIBILITY:
Key Inclusion Criteria:

* Patients who had low- and Int-1-risk myelodysplastic syndrome
* Documented diagnosis of the following:

Myelodysplastic syndrome that lasted ≥ 3 months and < 3 years Disease must not have been secondary to treatment with radiotherapy, chemotherapy, and/or immunotherapy for malignant or autoimmune diseases

* A hemoglobin < 10 g/dL and ≥ 8 g/dL
* History of transfusions < 10 RBC units and must not have been RBC transfusion dependent
* 300 ng/mL < serum ferritin < 1,500 ng/mL (Values within 10% difference above 1500 ng/ml or 10% difference below 300 ng/ml could have been accepted at the investigator's discretion.
* Endogenous erythropoietin levels < 500 units/L
* Serum creatinine ≤ 1.5 times upper limit of normal (ULN)
* Creatinine clearance above the concentration limit in locally approved prescribing information (PI). Patients with creatinine clearance between 40 and less than 60 mL/min, who did not present with additional risk factors that might impair renal function, were eligible at the discretion of the investigator

Key Exclusion Criteria:

* Patients who had MDS with isolated del(5q)
* Patients who had received prior EPO treatment or other recombinant growth factors regardless of the outcome (Patient who had received prior EPO treatment or other recombinant growth factors for less than 4 weeks and not within 3 months before screening without a documented response are allowed)
* Patients who had received steroids or immunosuppressive therapy for the improvement of hematological parameters (stable steroid treatment for adrenal failure or chronic medical conditions, and intermittent dexamethasone as antiemetics were allowed).
* B12 and folate deficient patients with and without clinical symptoms (patients were rescreened after successful therapy of B12 and folate deficiency)
* Uncontrolled seizures or uncontrolled hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-01-28 (Actual); Primary Completion 2017-03-22 (Actual); Study Completion 2017-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (30):
- Algeria (2):
  - Novartis Investigative Site, Oran
  - Novartis Investigative Site, Sidi Bel Abbes
- Argentina (2):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, La Plata, Buenos Aires
- Canada (3):
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, Toronto, Ontario
- China (6):
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Shanghai
- Germany (5):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Lütten Klein
  - Novartis Investigative Site, Würzburg
- Italy (3):
  - Novartis Investigative Site, Cagliari, CA
  - Novartis Investigative Site, Reggio Calabria, RC
  - Novartis Investigative Site, Roma, RM
- Novartis Investigative Site, Seoul, Korea, South Korea
- Spain (3):
  - Novartis Investigative Site, Badalona, Catalonia
  - Novartis Investigative Site, Girona, Catalonia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia
- Sweden (4):
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Linköping
  - Novartis Investigative Site, Luleå
  - Novartis Investigative Site, Stockholm
- Novartis Investigative Site, Oldham, Lancashire, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Twenty-three patients were randomized into the trial
Groups:
- Erythropoietin Alpha: Starting dose was erythropoietin 40,000 units/week. If after 4 weeks erythroid improvement was inadequate, dose was escalated to 60,000 units/week. If after 12 weeks of treatment, erythroid improvement was inadequate, participants were switched to the combination arm. At any time when erythroid response was achieved, erythropoietin treatment was stopped until end of study.
- Deferasirox + Erythropoietin Alpha: Starting dose was deferasirox dispersible tablet (DT) 10 mg/kg/day or deferasirox film-coated tablet FCT) 7 mg/kg/day in combination with erythropoietin 40,000 units/week. If after 4 weeks erythroid improvement was inadequate, erythropoietin dose was escalated to 60,000 units/week. If after 12 weeks of treatment, erythroid improvement was inadequate, participants were discontinued from the study. At any time when erythroid response was achieved, erythropoietin treatment was stopped study and Deferasirox treatment was continued until end of study
Period: Overall Study
Arm/Group | Erythropoietin Alpha | Deferasirox + Erythropoietin Alpha
Started | 12 | 11
Switched to EPO+DFX (Non-responders who switched to combination therapy at 12 weeks) | 5 | 0
Not Switched to EPO+DFX (Responders who were not switched to combination therapy at 12 weeks) | 7 | 0
Completed | 8 | 6
Not Completed | 4 | 5
Not completed — Adverse Event | 2 | 4
Not completed — Disease progression | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Erythropoietin Alpha | Deferasirox + Erythropoietin Alpha | Total
Number analyzed (Participants) | 12 | 11 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.5 (5.84) | 71.1 (7.54) | 72.9 (6.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 4 | 6 | 10
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 8 | 7 | 15
  Asian | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Difference in Percentage of Patients Achieving Erythroid Response Within 12 Weeks, by Treatment Group (Full Analysis Set)
Description: Difference in percentage of patients achieving an erythroid response within 12 weeks of treatment between the two arms according to modified IWG 2006 criteria increase in hemoglobin (Hb) ≥ 1.5 g/dL. Erythroid response is defined as the increase in Hb from baseline ≥ 1.5 g/dL. Patients achieving erythroid response at least once within 12 weeks were considered responders
Time Frame: Baseline up to 12 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Erythropoietin Alpha | Deferasirox + Erythropoietin Alpha
Number analyzed (Participants) | 12 | 11
percentage of participants | 41.7 [15.2 to 72.3] | 27.3 [6.02 to 61.0]
Statistical Analysis 1: Comparison: Erythropoietin Alpha vs Deferasirox + Erythropoietin Alpha; Test type: Other — difference; Mean Difference (Final Values) = 14.4, 95% CI 2-sided [-24.0 to 48.16]

2. Secondary Outcome: Absolute Change From Baseline to Post-baseline Value for Hemoglobin(g/dL)(Full Analysis Set)
Description: Hematological response criteria defined as: Erythroid response: hemoglobin (Hb) increase from baseline >= 1.5 g/dL (baseline < 11 g/dL), neutrophil response: increase from baseline >= 100% and increase > 0.5 × 10^9/L (baseline <1 × 10^9/L), platelet response: increase from baseline >= 30 × 10^9/L (baseline <100 × 10^9/L) according to modified IWG 2006 criteria
Time Frame: Baseline up to 24 weeks
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Erythropoietin Alpha | Deferasirox + Erythropoietin Alpha
Number analyzed (Participants) | 12 | 11
g/dL | 1.8 (0.21) | 2.1 (0.61)

3. Secondary Outcome: Summary of Hematologic Improvement in Patients Randomized to EPO+DFX and EPO Alone, Within 24 Weeks of Treatment (Full Analysis Set)
Description: Percentage of participants achieving an hematologic improvement defined as: neutrophil improvement: increase from baseline >0.5 × 10^9/L (baseline = 1.0 × 10^9/L ), platelet improvement: increase from baseline ≥ 30 × 10^9/L (baseline = 100 × 10^9/L), hemoglobin improvement: Hb increase from baseline ≥ 1 g/dL (baseline<11 g/dL)
Time Frame: Baseline up to 24 weeks
Population: Number of patients who met criteria varied across parameters
Measure: Number; unit: percentage of participants
Arm/Group | Erythropoietin Alpha | Deferasirox + Erythropoietin Alpha
Number analyzed (Participants) | 12 | 11
percentage of participants
  Hematologic improvement: number analyzed (Participants) | 12 | 5
  Hematologic improvement | 100 | 45.5
  Neutropil improvement: number analyzed (Participants) | 8 | 4
  Neutropil improvement | 66.7 | 80.0
  Platelet improvement: number analyzed (Participants) | 6 | 4
  Platelet improvement | 50.0 | 80.0
  Hemoglobin improvement: number analyzed (Participants) | 8 | 3
  Hemoglobin improvement | 66.7 | 60.0

4. Secondary Outcome: Absolute Change in Hemoglobin Values up to 24 Weeks
Description: Absolute change in hemoglobin values for patients showing improvement: Hemoglobin improvement Hb increase from baseline ≥ 1 g/dL (baseline<11 g/dL)
Time Frame: Baseline up to 24 weeks
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Erythropoietin Alpha | Deferasirox + Erythropoietin Alpha
Number analyzed (Participants) | 12 | 11
g/dL | 1.3 (0.37) | 1.4 (0.55)

5. Secondary Outcome: Absolute Change in Platelets and Neutrophil Levels up to 24 Weeks
Description: Absolute change in platelets and neutrophil levels for participants showing improvement: neutrophil improvement: increase from baseline >0.5 × 10^9/L (baseline = 1.0 × 10^9/L ), platelet improvement: increase from baseline ≥ 30 × 10^9/L (baseline = 100 × 10^9/L)
Time Frame: Baseline up to 24 weeks
Population: Number of patients who met criteria varied across parameters
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Erythropoietin Alpha | Deferasirox + Erythropoietin Alpha
Number analyzed (Participants) | 12 | 11
10^9 cells/L
  Platelets: number analyzed (Participants) | 6 | 4
  Platelets | 58.7 (23.93) | 66.3 (22.74)
  Neutrophils: number analyzed (Participants) | 8 | 4
  Neutrophils | 1.2 (1.16) | 2.4 (1.57)

6. Secondary Outcome: Summary of Erythroid Response in Participants Randomized to EPO Alone at Baseline and Switched to EPO+DFX After 12 Weeks of Treatment (Full Analysis Set)
Description: Erythroid response: hemoglobin increase from baseline > = 1.5 g/dL (baseline <11 g/dL)
Time Frame: Week 13 up to 24 weeks
Measure: Number; unit: participants
Groups:
- EPO+DFX (12 Weeks): Patients randomized to EPO alone with inadequate response at 12 weeks who had been switched over to combination EPO+DFX
Arm/Group | EPO+DFX (12 Weeks)
Number analyzed (Participants) | 5
participants | 0

7. Secondary Outcome: Summary of Erythroid Response Within 24 Weeks in Participants Randomized to EPO at Baseline and Not Switched to EPO+DFX After 12 Weeks of Treatment (Full Analysis Set)
Description: Erythroid response: hemoglobin increase from baseline > = 1.5 g/dL (baseline <11 g/dL). Percentages are based on N. Confidence intervals are calculated using Clopper-Pearson method. Hemoglobin value is at time of first response
Time Frame: baseline up to 24 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- EPO (24 Weeks): Patients who were in EPO alone group and were not switched to EPO+DFX after 12 weeks,
Arm/Group | EPO (24 Weeks)
Number analyzed (Participants) | 7
percentage of participants | 71.4 [47.8 to 100.0]

8. Secondary Outcome: Absolute Change in Serum Ferritin up to 24 Weeks for Erythropoietin Alpha Arm (Full Analysis Set)
Description: Absolute change in serum ferritin from baseline
Time Frame: Baseline up to 24 weeks
Population: Number of patients analyzed varied by visit
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Erythropoietin Alpha
Number analyzed (Participants) | 7
ng/mL
  Responders - Week 5: number analyzed (Participants) | 5
  Responders - Week 5 | -98.5 [-323 to -73.5]
  Responders - Week 9: number analyzed (Participants) | 5
  Responders - Week 9 | -79.0 [-381 to 54.0]
  Responders - Week 13: number analyzed (Participants) | 4
  Responders - Week 13 | 24.8 [-179 to 104]
  Responders - Week 17: number analyzed (Participants) | 4
  Responders - Week 17 | -57.8 [-140 to 258.0]
  Responders - Week 21: number analyzed (Participants) | 2
  Responders - Week 21 | -39.8 [-44.0 to -35.5]
  Non-responders - Week 5: number analyzed (Participants) | 2
  Non-responders - Week 5 | -352 [-523 to -182]
  Non-responders - Week 9: number analyzed (Participants) | 2
  Non-responders - Week 9 | -189 [-572 to 194.5]
  Non-responders - Week 13: number analyzed (Participants) | 2
  Non-responders - Week 13 | -44.5 [-621 to 531.5]

9. Secondary Outcome: Absolute Change in Serum Ferritin up to 24 Weeks for Deferasirox + Erythropoietin Alpha Arm (Full Analysis Set)
Description: Absolute change in serum ferritin from baseline
Time Frame: Baseline up to 24 weeks
Population: Number of patients analyzed varied by visit
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Deferasirox + Erythropoietin Alpha
Number analyzed (Participants) | 11
ng/mL
  Responders - Week 5: number analyzed (Participants) | 3
  Responders - Week 5 | -82.5 [-243 to 1068]
  Responders - Week 9: number analyzed (Participants) | 3
  Responders - Week 9 | -139 [-292 to 702.0]
  Responders - Week 13|: number analyzed (Participants) | 3
  Responders - Week 13| | -121 [-338 to 0.0]
  Responders - Week 17: number analyzed (Participants) | 3
  Responders - Week 17 | 16.5 [-143 to 722.0]
  Responders - Week 21: number analyzed (Participants) | 3
  Responders - Week 21 | -95.5 [-189 to 173.0]
  Non-responders - Week 5: number analyzed (Participants) | 7
  Non-responders - Week 5 | -38.0 [-315 to 111.0]
  Non-responders - Week 9|: number analyzed (Participants) | 4
  Non-responders - Week 9| | -144 [-435 to 1.0]
  Non-responders - Week 13|: number analyzed (Participants) | 3
  Non-responders - Week 13| | -155 [-225 to -127]
  Non-responders - Week 17: number analyzed (Participants) | 2
  Non-responders - Week 17 | -123 [-154 to -91.0]
  Non-responders - Week 21: number analyzed (Participants) | 1
  Non-responders - Week 21 | -291 [-291 to -291]

10. Secondary Outcome: Absolute Change in Serum Ferritin up to 24 Weeks for EPO+DFX at 12 Weeks Arm (Full Analysis Set)
Description: Absolute change in serum ferritin from baseline
Time Frame: Baseline up 24 weeks
Population: Number of patients analyzed varied by visit
Measure: Median (Full Range); unit: ng/mL
Groups:
- EPO+DFX at 12: Patients randomized to EPO alone with inadequate response at 12 weeks who had been switched over to combination EPO+DFX
Arm/Group | EPO+DFX at 12
Number analyzed (Participants) | 5
ng/mL
  Responders - Week 5: number analyzed (Participants) | 1
  Responders - Week 5 | -116 [-116 to -116]
  Responders - Week 9: number analyzed (Participants) | 1
  Responders - Week 9 | -136 [-136 to -136]
  Responders - Week 13: number analyzed (Participants) | 1
  Responders - Week 13 | 59.5 [59.5 to 59.5]
  Responders - Week 17: number analyzed (Participants) | 1
  Responders - Week 17 | 74.5 [74.5 to 74.5]
  Non-responders - Week 5: number analyzed (Participants) | 4
  Non-responders - Week 5 | -68.3 [-144 to 221.3]
  Non-responders - Week 9: number analyzed (Participants) | 3
  Non-responders - Week 9 | -148 [-319 to 321.3]
  Non-responders - Week 13: number analyzed (Participants) | 4
  Non-responders - Week 13 | 220.4 [-228 to 635.3]
  Non-responders - Week 17: number analyzed (Participants) | 2
  Non-responders - Week 17 | -16.6 [-28.5 to -4.7]
  Non-responders - Week 21: number analyzed (Participants) | 3
  Non-responders - Week 21 | -10.5 [-463 to 367.3]

11. Secondary Outcome: Absolute Change in Hemoglobin (Hb) From Baseline for Erythropoietin Alpha Arm (Full Analysis Set)
Description: This analysis included patients randomized either to EPO or DFX+EPO at baseline as well as patients who did not have erythroid response at week 12 in the EPO group and switched to combination therapy.
Time Frame: Baseline up to 24 weeks
Population: Number of patients analyzed varied by visit
Measure: Median (Full Range); unit: g/dL
Arm/Group | Erythropoietin Alpha
Number analyzed (Participants) | 7
g/dL
  Responders - Week 5: number analyzed (Participants) | 5
  Responders - Week 5 | 1.5 [1.1 to 3.2]
  Responders - Week 9: number analyzed (Participants) | 5
  Responders - Week 9 | 1.9 [1.3 to 4.4]
  Responders - Week 13: number analyzed (Participants) | 4
  Responders - Week 13 | 1.7 [1.5 to 3.4]
  Responders - Week 17: number analyzed (Participants) | 4
  Responders - Week 17 | 1.6 [-0.3 to 1.8]
  Responders - Week 21: number analyzed (Participants) | 3
  Responders - Week 21 | 0.8 [-0.7 to 1.8]
  Non-responders - Week 5: number analyzed (Participants) | 2
  Non-responders - Week 5 | -0.9 [-1.7 to -0.1]
  Non-responders - Week 9: number analyzed (Participants) | 2
  Non-responders - Week 9 | -1.7 [-2.0 to -1.4]
  Non-responders - Week 13: number analyzed (Participants) | 2
  Non-responders - Week 13 | -2.5 [-2.8 to -2.1]

12. Secondary Outcome: Absolute Change in Hemoglobin (Hb) From Baseline for Deferasirox + Erythropoietin Alpha Arm (Full Analysis Set)
Description: as for outcome 11
Time Frame: Baseline up to 24 weeks
Population: Number of patients analyzed varied by visit
Measure: Median (Full Range); unit: g/dL
Arm/Group | Deferasirox + Erythropoietin Alpha
Number analyzed (Participants) | 11
g/dL
  Responders - Week 5: number analyzed (Participants) | 3
  Responders - Week 5 | 0.7 [0.6 to 2.0]
  Responders - Week 9: number analyzed (Participants) | 3
  Responders - Week 9 | 1.6 [1.0 to 2.6]
  Responders - Week 13: number analyzed (Participants) | 3
  Responders - Week 13 | 2.9 [2.8 to 3.0]
  Responders - Week 17: number analyzed (Participants) | 3
  Responders - Week 17 | 2.4 [0.6 to 3.0]
  Responders - Week 21: number analyzed (Participants) | 3
  Responders - Week 21 | 1.7 [-1.3 to 2.4]
  Non-responders - Week 5: number analyzed (Participants) | 7
  Non-responders - Week 5 | -0.1 [-2.3 to 0.1]
  Non-responders - Week 9: number analyzed (Participants) | 4
  Non-responders - Week 9 | 0.0 [-0.8 to 0.5]
  Non-responders - Week 13: number analyzed (Participants) | 3
  Non-responders - Week 13 | 0.2 [0.1 to 0.5]
  Non-responders - Week 17: number analyzed (Participants) | 1
  Non-responders - Week 17 | -0.5 [-0.5 to -0.5]
  Non-responders - Week 21: number analyzed (Participants) | 1
  Non-responders - Week 21 | -0.6 [-0.6 to -0.6]

13. Secondary Outcome: Absolute Change in Hemoglobin (Hb) From Baseline for EPO+DFX at 12 Weeks Arm (Full Analysis Set)
Description: This analysis included patients randomized either to EPO or DFX+EPO at baseline as well as patients who did not have erythroid response at week 12 in the EPO group and switched to combination therapy. The time-course of Hb and its absolute changes from baseline was summarized by descriptive statistics by visit and erythroid response. Patients randomized to EPO and not switching after 12 weeks to EPO+DFX would consist of only responders.
Time Frame: Baseline up to 24 weeks
Population: Number of patients analyzed varied by visit
Measure: Median (Full Range); unit: g/dL
Groups:
- EPO+DFX at 12 Weeks: This analysis included patients randomized either to EPO or DFX+EPO at baseline as well as patients who did not have erythroid response at week 12 in the EPO group and switched to combination therapy. The time-course of Hb and its absolute changes from baseline was summarized by descriptive statistics by visit and erythroid response. Patients randomized to EPO and not switching after 12 weeks to EPO+DFX would consist of only responders
Arm/Group | EPO+DFX at 12 Weeks
Number analyzed (Participants) | 5
g/dL
  Responders - Week 5: number analyzed (Participants) | 1
  Responders - Week 5 | 1.2 [1.2 to 1.2]
  Responders - Week 9|: number analyzed (Participants) | 1
  Responders - Week 9| | 1.8 [1.8 to 1.8]
  Responders - Week 13|: number analyzed (Participants) | 1
  Responders - Week 13| | 0.7 [0.7 to 0.7]
  Responders - Week 17|: number analyzed (Participants) | 1
  Responders - Week 17| | -0.6 [-0.6 to -0.6]
  Non-responders - Week 5: number analyzed (Participants) | 4
  Non-responders - Week 5 | 0.3 [-0.5 to 0.6]
  Non-responders - Week 9|: number analyzed (Participants) | 3
  Non-responders - Week 9| | 0.5 [-0.4 to 0.8]
  Non-responders - Week 13: number analyzed (Participants) | 3
  Non-responders - Week 13 | 0.4 [0.2 to 1.0]
  Non-responders - Week 17|: number analyzed (Participants) | 3
  Non-responders - Week 17| | 0.0 [-0.1 to 0.9]
  Non-responders - Week 21: number analyzed (Participants) | 3
  Non-responders - Week 21 | 0.0 [-0.7 to 0.8]

ADVERSE EVENTS:
Time Frame: Adverse Events are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All Adverse events are reported in this record from First Patient First Treatment until Last Patient Last Visit up to approximately 24 weeks
Description: There was no washout period during the study before switch of treatment. Therefore effects (including AEs) from long lasting treatment like EPO can potentially still be observed after the switch, e.g. from EPO+DFX to DFX alone. Thus the resulting includes both treatments (DFX-EPO category). The same applies for staring EPO alone and switching to EPO plus DFX.
Groups:
- EPO A: Patients receiving EPO during the first 12 weeks and no switching to EPO+DFX arm
- EPO+DFX DT: Patients receiving EPO+DFX from week 1 and continuing with EPO+DFX after 12 weeks or with DFX alone after 12 weeks
- EPO+DFX FCT: Patients receiving EPO alone and switched to EPO+DFX after 12 weeks of treatment
- Switched to DFX+EPO After 12 Weeks: Switched to DFX+EPO after 12 weeks
Arm/Group | EPO A | EPO+DFX DT | EPO+DFX FCT | Switched to DFX+EPO After 12 Weeks
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/10 | 0/1 | 0/5
Serious Adverse Events (participants affected / at risk) | 1/7 | 1/10 | 1/1 | 1/5
Other Adverse Events (participants affected / at risk) | 4/7 | 10/10 | 1/1 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EPO A (N=7) | EPO+DFX DT (N=10) | EPO+DFX FCT (N=1) | Switched to DFX+EPO After 12 Weeks (N=5)
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
C-reactive protein increased (Investigations) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | EPO A (N=7) | EPO+DFX DT (N=10) | EPO+DFX FCT (N=1) | Switched to DFX+EPO After 12 Weeks (N=5)
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Anal fissure (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 1 | 0 | 0
Gravitational oedema (General disorders) | 0 | 1 | 0 | 0
Injection site bruising (General disorders) | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 2
Lung infection (Infections and infestations) | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 0 | 0
Heart rate increased (Investigations) | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2015-08-06): https://cdn.clinicaltrials.gov/large-docs/77/NCT01868477/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-12): https://cdn.clinicaltrials.gov/large-docs/77/NCT01868477/SAP_001.pdf